CLINICAL TRIAL: NCT02928796
Title: Attentional Capacity and Clinician Performance: Eye-Tracking Participants When Using a High-Fidelity Surgical Simulator That Emulates Cardiology Procedures
Brief Title: Attentional Capacity and Clinician Performance
Acronym: ACCP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Principal Investigator, Prof Anthony G. Gallagher, Director of Research, Professor of Technology Enhanced Learning, University College Cork
Other Study IDs: ACCP - 1
Record Dates: First submitted 2016-09-30; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Change in Sustained Attention
Keywords: Attentional capacity; Working memory; Simulation-based training; Eye-tracking; Visual attention; Psychophysiological measurement; Surgical simulation; Computer-based simulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Trainees: Registrar Cardiologists
  Interventions: Behavioral: Cognitive Stimulus
- Trainers: Consultant Cardiologists
  Interventions: Behavioral: Cognitive Stimulus

INTERVENTIONS:
Behavioral: Cognitive Stimulus — Participants to pay attention to a supplementary display monitor and respond to specified stimulus images, all while performing the simulated cardiology-based procedure.

SUMMARY:
Uncovering the distinct measurements and features that potentially exist in different levels of expertise when performing cardiology-based procedures. There is a belief that tracking the visual attention and other psychophysiological measures during performance of these procedures may assist in uncovering the attentional capacity of participants and how it links with overall performance.

DETAILED DESCRIPTION:
Attentional capacity is the number of items a person can hold in their temporal memory whilst undertaking a task (researchers equivocate this to Random Access Memory in computing hardware). Therefore, attentional capacity is thought to play a role in task performance and if a person's attentional capacity is measured 'in-vivo' then one can predict that person's ability and aptitude (classifying if they are an expert or novice since an expert will not require the full capacity of their temporal capacity, as many of the routine steps are stored in their permanent memory). The measurement of performance is of interest in medical training and competency testing research. Eye-tracking and other novel methods could offer new and effective components for measuring performance during complex procedures. These novel methods have increasingly been spotted in new healthcare research studies which aim to use them for a multitude of purposes, mostly to uncover valuable insights between different participant performance levels. One form of medical training is high-fidelity virtual reality simulators that can provide an almost life-like training environment for the trainee and one common use of these simulators is for surgical training . Some work with eye-tracking has already been done with surgical tasks that indicates visual attention does discriminate between novice and expert level performance. There is scope for using eye-tracking technology to capture visual attention during complex surgical procedures to uncover the discriminatory measurements between participants at different levels of expertise.

Aims The first aim of the study is to investigate the relationship between attentional capacity and performance during cardiology-based procedures. The hypothesise is that a significant relationship will be found and that attentional capacity will be a statistically significant predictor for discriminating between experts and novices.

The second aim of the study is to investigate the relationship between visual attention (recorded via eye tracking) and the precisely recorded actions taken by the participant during the procedure.

A third aim of the study is to investigate the relationship between physiological metrics (Heart rate, GSR recorded via E4 wristband) and the precisely recorded actions taken by the participant during the procedure.

This will be facilitated by the capture of the participant's visual attention, through worn eye-tracking glasses, level of arousal, through worn GSR/EDA wristband and their verbalisation (thinking-aloud during task performance), recorded through video/microphone, during two simulated cardiology-based procedures. The simulator will provide its own metrics (duration etc.) to represent the participants' performance during the procedure. The simulation will be provided by a state of the art of surgical simulator in the ASSERT Centre, University College Cork. An extra display monitor will also be included to provide the extra stimulus to assess attentional capacity. The monitor will display a specific playing card at certain times during the proceedings. The participant will have to acknowledge what the card was. This and the visual attention capture will provide insight to the participants' attentional capacity.

ELIGIBILITY:
Inclusion Criteria:

* They must be qualified medical doctor with specific interest in cardiology (e.g. consultant cardiologist). Consultant group must contain consultants only and registrar group must have enrolled registrars only.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Qualified medical professionals, trainees/registrars or trainers/consultants, working within the cathlab environment and discipline of interventional cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Mean attentional capacity | Up to 12 Months.
  The hypothesis is that a significant statistical relationship will be found between measured attentional capacity (via a card reading task) and overall surgical task performance grading. Attentional capacity, we hypothesise, will be a statistically significant predictor for discriminating between performance level.
Visual attention characteristics for stimulus reading 'card' task | Up to 12 months.
  The hypothesis is that a significant statistical relationship will be found with characteristics of participant's visual attention (e.g. mean fixation duration, mean saccade latency, overall visual latency before card acknowledgement) and the measured attentional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony G. Gallagher, DSc, PhD, Principal Investigator — University College Cork
Locations (1):
- ASSERT Centre, University College Cork, Cork, Cork, Ireland

REFERENCES:
- [Derived] Currie J, Bond RR, McCullagh P, Black P, Finlay DD, Gallagher S, Kearney P, Peace A, Stoyanov D, Bicknell CD, Leslie S, Gallagher AG. Wearable technology-based metrics for predicting operator performance during cardiac catheterisation. Int J Comput Assist Radiol Surg. 2019 Apr;14(4):645-657. doi: 10.1007/s11548-019-01918-0. Epub 2019 Feb 7. PMID 30730031